CLINICAL TRIAL: NCT04518085
Title: Pre- and Post-operative Psychological Interventions to Prevent Pain and Fatigue After Breast Cancer Surgery: a Randomized Controlled Trial
Brief Title: Psychological Interventions to Prevent Late Effects in Breast Cancer
Acronym: PREVENT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oslo (Other)
Collaborators: Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Silje Endresen Reme, Professor, University of Oslo
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 201906
Record Dates: First submitted 2020-08-05; First posted 2020-08-19 (Actual); Last update posted 2023-12-08 (Actual); Status verified 2023-12

CONDITIONS: Pain, Postoperative; Fatigue; Breast Cancer
Keywords: Breast cancer; Post-surgical pain; Fatigue; Hypnosis; Acceptance and commitment therapy
MeSH Terms: conditions — Pain, Postoperative; Fatigue; Breast Neoplasms | interventions — Therapeutics

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial, in which participants are randomly allocated to either the intervention group or an active control group.
Who Masked: Investigator, Outcomes Assessor
Masking Description: The intervention group vs. active control group status will be known to the participants and the health care personnel delivering the interventions. However, the investigator, outcome assessor and the additional health care personnel at the unit will be masked to the conditions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hypnosis + iACT (Experimental): Single 20 minute medical hypnosis session delivered pre-surgery plus internet-based acceptance and commitment therapy delivered post-surgery
  Interventions: Behavioral: Medical hypnosis; Behavioral: Internet-based Acceptance and Commitment Therapy (iACT)
- Mindfulness + treatment as usual (TAU) (Active Comparator): Single 20 minute mindfulness session delivered pre-surgery plus treatment as usual post-surgery
  Interventions: Behavioral: Mindfulness session; Behavioral: Treatment as Usual (TAU)

INTERVENTIONS:
Behavioral: Medical hypnosis — Single session 20 minutes hypnosis session originally developed and tested by Montgomery et al. (2007) in a similar setting. Delivered by an experienced clinical psychologist.
  Arms: Hypnosis + iACT
Behavioral: Internet-based Acceptance and Commitment Therapy (iACT) — Access to an online platform developed to this study containing video clips and audio files with ACT consistent material
  Arms: Hypnosis + iACT
Behavioral: Mindfulness session — Single session mindfulness session delivered by audio file
  Arms: Mindfulness + treatment as usual (TAU)
Behavioral: Treatment as Usual (TAU) — Treatment as usual as part of post-surical care
  Arms: Mindfulness + treatment as usual (TAU)

SUMMARY:
The study aims to investigate whether a combined pre-operative medical hypnosis plus a post-operative internet-based acceptance and commitment intervention are more effective in preventing post-surgical pain and fatigue following breast cancer surgery compared with pre-operative mindfulness plus treatment as usual.

DETAILED DESCRIPTION:
The trial will include 200 patients undergoing breast cancer surgery at Oslo University Hospital. The patients will be randomized into two groups. One group will receive a 20 minute pre-surgical hypnosis session delivered by an experienced clinical psychologist plus a post-surgical internet-based acceptance and commitment intervention. The control group will receive a 20 minute pre-surgical mindfulness session delivered through an audio recording plus treatment as usual. The primary outcomes of the study are quantitative measures of post-surgical pain and fatigue. In addition, relationships between biomarkers of stress and subacute post-surgical pain and fatigue will be analyzed using using blood- and hair samples. The study uses a longitudinal design with baseline measures obtained pre-surgery and follow up measures obtained 3 and 12 months post-surgery.

ELIGIBILITY:
Inclusion Criteria:

* Women diagnosed with breast cancer and scheduled for surgery
* Be able to provide informed consent

Exclusion Criteria:

* Insufficient Norwegian speaking or writing skills to participate in the interventions and fill out questionnaires
* Cognitive and psychiatric impairment
* Other serious malignancies

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Eligible participants are women (biological sex) diagnosed with breast cancer
Enrollment: 203 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2022-03-03 (Actual); Study Completion 2023-11-01 (Actual)

PRIMARY OUTCOMES:
Chronic post-surgical pain | 3 months after surgery
  Measured through a Numeric Rating Scale (NRS) for pain intensity. The scale ranges from 0-10, anchored by verbal descriptors at either end of the scale where 0 is no pain at all and 10 is the worst possible pain.
Post-surgical fatigue | 3 months after surgery
  Measured through the 13-item Functional Assessment of Chronic Illness Therapy-Fatigue subscale (FACIT-F) which is a unidimensional self-report scale to assess fatigue and its impact on daily life. The score range is 0-52 where a higher score indicates better quality of life (i.e. less symptoms and disability)

SECONDARY OUTCOMES:
Pain intensity, pain unpleasantness, fatigue, nausea, physical discomfort and emotional upset | On the day of surgery right before discharge
  Measured by a Visual Analogue Scale (VAS) (to replicate a previous hypnosis trial - Montgomery et al 2007). The range is 0-100 where a higher score indicates more intense symptoms.
Stress (immunological) reactivity | Baseline (pre-surgery) plus 4 weeks post-surgery (Cortisol will only be measured at baseline)
  Immune function is assessed through whole blood samples using the standardized TruCulture system that contains immunogenic stimuli (infected tubes). This test will reveal the induced innate and adaptive immune response in whole blood after stimulation with LPS, by quantifying the release of soluble immune activation products (cytokines, chemokines, soluble receptors etc.) in the supernatant and by measuring the transcription level (mRNA) in the circulating blood (immune) cells.
Number of psychotropic and pain-related prescriptions | 3 and 12 months post-surgery
  Usage of psychotropic and pain medication obtained through registry data from the Norwegian Prescription Database at 3 and 12 months follow-up. Number of prescriptions will be summarized and compared between intervention and control group.
Number of sick leave days | 3 and 12 months post-surgery
  Days away from work on sick leave will be measured through registry data
Psychological flexibility | 3 and 12 months post-surgery
  Measured through the Acceptance and Action Questionnaire (AAQ-II). The scale ranges from 7-49, where higher score indicates more psychological inflexibility
Psychological distress | 3 and 12 months post-surgery
  Measured through the Hospital Anxiety and Depression Scale (HADS). The total score ranges from 0-42, where a higher score indicates more symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Silje E Reme, PhD, Principal Investigator — University of Oslo + Oslo University Hospital; Henrik B Jacobsen, PhD, Principal Investigator — University of Oslo + Oslo University Hospital
Locations (1):
- Oslo University Hospital (Aker Hospital), Oslo, Norway

IPD SHARING:
Plan to Share IPD: Yes
The study protocol, along with the intervention protocols, will all be published and publicly available. Registry data will not be shared as this is not allowed to share according to Norwegian law. However, data files involving questionnaire and biomarker data will be made available upon reasonable request. Due to privacy concerns, the complete data files will not be shared online.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: The study protocol will be published as soon as possible. The intervention protocols will be publicly available upon study completion. Data files will be made available when the main analyses are completed, in 2025 at the latest.
Access Criteria: Data files involving self-report data will be shared upon reasonable request when the main analyses are completed and published.

REFERENCES:
- [Background] Lind SB, Jacobsen HB, Solbakken OA, Reme SE. Clinical Hypnosis in Medical Care: A Mixed-Method Feasibility Study. Integr Cancer Ther. 2021 Jan-Dec;20:15347354211058678. doi: 10.1177/15347354211058678. PMID 34818921
- [Background] Engel S, Jacobsen HB, Reme SE. A cross-sectional study of fear of surgery in female breast cancer patients: Prevalence, severity, and sources, as well as relevant differences among patients experiencing high, moderate, and low fear of surgery. PLoS One. 2023 Jun 23;18(6):e0287641. doi: 10.1371/journal.pone.0287641. eCollection 2023. PMID 37352256
- [Background] Munk A, Jacobsen HB, Schnur J, Montgomery G, Reme SE. Acute and subacute postsurgical pain in women with breast cancer: incidence and associations with biopsychosocial predictors-a secondary analysis of a randomized controlled trial. Pain Rep. 2023 Jan 10;8(1):e1058. doi: 10.1097/PR9.0000000000001058. eCollection 2023 Jan. PMID 36699993
- [Background] Reme SE, Munk A, Holter MTS, Falk RS, Jacobsen HB. Pre- and post-operative psychological interventions to prevent pain and fatigue after breast cancer surgery (PREVENT): Protocol for a randomized controlled trial. PLoS One. 2022 Jul 8;17(7):e0268606. doi: 10.1371/journal.pone.0268606. eCollection 2022. PMID 35802618
- [Derived] Reme SE, Munk A, Montgomery GH, Schnur JB, Falk R, Smits M, Jacobsen HB. Preoperative Hypnosis versus Mindfulness for Reducing Postoperative Symptoms in Breast Surgery: A Randomized Clinical Trial. Anesthesiology. 2026 Mar 1;144(3):559-569. doi: 10.1097/ALN.0000000000005821. Epub 2025 Nov 7. PMID 41203018
- See also: Project web page — https://www.sv.uio.no/psi/english/research/projects/pre-and-post-operative-psychological-interventions/index.html